CLINICAL TRIAL: NCT04086082
Title: MAGIK: Using Implanted Markers to Determine the Feasibility of Markerless Image Guidance Using Intrafraction Kilovoltage X-ray Imaging: A Phase I Interventional Study of Lung Cancer Radiotherapy
Brief Title: Markerless Image Guidance Using Intrafraction Kilovoltage X-ray Imaging
Acronym: MAGIK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAGIK V1.0
Record Dates: First submitted 2019-05-06; First posted 2019-09-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; NSCLC; Oligometastases
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Markerless Image Guidance Arm (Experimental): Single arm trial using implanted markers to determine the feasibility of Markerless Image Guidance using Intrafraction Kilovoltage X-ray Imaging
  Interventions: Device: Markerless Image Guidance

INTERVENTIONS:
Device: Markerless Image Guidance — Single arm trial using implanted markers to determine the feasibility of Markerless Image Guidance using Intrafraction Kilovoltage X-ray Imaging

SUMMARY:
This trial will investigate the feasibility of the Markerless Tumour Tracking technology.

DETAILED DESCRIPTION:
Markerless Tumour Tracking will be integrated with existing treatment machines to provide real-time monitoring of tumour motion during treatment delivery. Eligible patients will be implanted with fiducial markers, which act as the ground truth for evaluating the accuracy of Markerless Tumour Tracking. The patients will undergo the current standard of care radiotherapy, with the exception that kilovoltage x-ray images will be acquired continuously during treatment delivery to enable Markerless Tumour Tracking.

ELIGIBILITY:
Inclusion Criteria:

* Is willing to comply with all trial procedures and intends to provide written Informed Consent for participation in this trial.
* Patients undergoing external beam radiotherapy.
* Histologically proven Stage I NSCLC or oligometastatic lung metastases (3 or less).
* MRI/4D-CT prior to insertion of fiducial markers.
* Patient must be able to have fiducial markers placed in the lung (if on anticoagulants, must be cleared by LMO or cardiologist).
* ECOG performance status 0-2.
* A maximum of three metastases to the lung from any non-haematological malignancy. Multiple metastases will be treated separately.
* 1 cm ≤ Tumour diameter in any dimension ≤ = 5 cm.
* The distance between the tumour centroid and the top end of the diaphragm is <=10 cm.

Exclusion Criteria:

* Patient has low respiratory performance as evaluated by the physicians.
* Previous high-dose thoracic radiotherapy.
* Less than one fiducial marker implanted in the lung.
* Fiducial markers are too far from the tumour centroid (>9 cm).
* Cytotoxic chemotherapy within 3 weeks of commencement of treatment, or concurrently with treatment. Hormonal manipulation agents are allowable (e.g. aromatase inhibitors, selective oestrogen receptor modulators, and gonadotropin releasing hormone receptor modulators).
* Targeted agents (such as sunitinib, bevacizumab and tarceva) within 7 days of commencement of treatment, or concurrently with treatment.
* Women who are pregnant or lactating.
* Unwilling or unable to complete quality of life questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Markerless Tumour Tracking is feasible for motion-adaptive lung cancer radiotherapy | 2 years
  This will be measured by 90% of the treatment fractions achieving:
  1. Continuous on-line tracking with no software failure;
  2. Agreement between markerless and marker-based tracking within 3 mm in each direction (left-right, superior-inferior, anterior-posterior) for at least 80% of the beam-on time as assessed in off-line analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, PhD, Principal Investigator — University of Sydney
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data and images will be made available for other scientific research.
Supporting Information: Study Protocol
Time Frame: Data will be made available following publication of the final analysis, and for a minimum of 2 years thereafter.
Access Criteria: Requests must be made to the original researchers for access to the data.

REFERENCES:
- [Derived] Mueller M, Booth J, Briggs A, Jayamanne D, Panettieri V, Senthi S, Shieh CC, Keall P. MArkerless image Guidance using Intrafraction Kilovoltage x-ray imaging (MAGIK): study protocol for a phase I interventional study for lung cancer radiotherapy. BMJ Open. 2022 Jan 20;12(1):e057135. doi: 10.1136/bmjopen-2021-057135. PMID 35058267